CLINICAL TRIAL: NCT02959216
Title: Sub-Symptom Aerobic Exercise Therapy to Improve Recovery From Acute Sport-Related Concussion: A Randomized Controlled Trial
Brief Title: Aerobic Exercise for Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University at Buffalo (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-012491
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Mild Traumatic Brain Injury; Acute Brain Injury; Brain Concussion
Keywords: Aerobic Exercise
MeSH Terms: conditions — Brain Concussion; Brain Injuries | interventions — Exercise; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Aerobic exercise participants will receive an exercise prescription based on their heart rate threshold (HRT) for symptom exacerbation during an initial treadmill test. Participants will be asked to exercise once a day up to 90% of their assigned HRT for a minimum of 20 minutes. Participants will wear a heart rate monitor to track their heart rate during aerobic exercise. The treatment will continue until the participant is recovered from his/her concussion, as determined by exercise tolerance and a normal symptom count and clinical examination.
  Interventions: Other: Aerobic Exercise
- Stretching Exercise (Placebo Comparator): Stretching exercise participants will receive a prescription to complete a standardized physical therapy stretching protocol once a day for approximately 20 minutes. Participants will wear a heart rate monitor to track their heart rate during the stretching exercise. The treatment will continue until the participant is recovered from his/her concussion, as determined by exercise tolerance and a normal symptom count and clinical examination.
  Interventions: Other: Stretching Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Participants will be given a prescription to exercise up to 90% of their threshold heart rate for symptom exacerbation. Heart rate threshold will be monitored weekly in order to increase exercise level accordingly.
  Arms: Aerobic Exercise
Other: Stretching Exercise — Participants will be given a prescription to complete a standardized stretching protocol.
  Arms: Stretching Exercise

SUMMARY:
The use of aerobic exercise treatment in the chronic phase of concussion recovery is well-described in the literature but there are limited existing data on the effect of exercise treatment in the acute phase after sport-related concussion (SRC). This study will compare the outcomes of adolescents with a recent SRC who are randomized to sub-threshold aerobic exercise versus those randomized to placebo stretching to evaluate the effect of aerobic exercise in the acute recovery phase.

DETAILED DESCRIPTION:
Historically, concussion has been described as a cognitive injury and patients have been advised not to engage in any cognitive or physical exertion while symptomatic. More recently, however, concussion has been described as a physiological injury affecting both the heart and autonomic nervous system, and patients suffering from prolonged concussion-related symptoms and deficits have been encouraged to begin aerobic exercise as part of their concussion care. While intensive exercise too soon after concussion has been associated with delayed recovery and used to justify prolonged periods of rest, recent studies have shown that controlled, sub-symptom threshold aerobic exercise may aid recovery by improving autonomic balance and cerebral blood flow auto-regulation after concussion. This study will randomly assign pediatric patients with concussion to a treatment group in which they will complete sub-symptom threshold aerobic exercise or to a placebo group in which they will complete a standardized stretching protocol. All participants will have routine visits that consist of a physical examination and exercise test until the intervention ends at recovery or 1-month post-randomization.

ELIGIBILITY:
Inclusion Criteria (Case Subjects):

* Sports-related concussion (organized or recreational).
* Physician-diagnosed concussion within the last 10 days.
* Symptom score difference ≥3 on the Post-Concussion Symptom Inventory (PCSI) Current versus PCSI Pre-Injury.
* Parental/guardian permission (informed consent) and child assent.

Inclusion Criteria (Control Subjects):

* No known recent concussion within the past year or still causing active symptoms.
* Parental/guardian permission (informed consent) and child assent.

Exclusion Criteria (Case and Control Subjects):

* Subjects with moderate or severe traumatic brain injury as indicated by a score <13 on Glasgow Coma Scale (GCS), presence of lesion on CT/MRI, and/or focal neurologic deficit consistent with an intracerebral lesion.
* History of more than 3 diagnosed concussions.
* Subjects that sustained an injury involving loss of consciousness for 30+ minutes or post-traumatic amnesia for 24+ hours.
* Inability to exercise because of lower-extremity orthopedic injury, significant vestibular or visual dysfunction, or increased cardiac risk.
* Pre-existing comorbidities, such as chronic pain, cardiac, neurological, or autoimmune conditions, that prevent participation in active testing and/or rehabilitation.
* Currently taking medications that can affect autonomic function.
* Active substance abuse/dependence.
* Unwillingness to exercise or unable to access place to safely exercise.
* Parental/guardian permission (informed consent) not obtainable or not provided
* Cannot understand English.

Exclusion Criteria (Case Subjects Only):

* Additional head injury during the intervention.
* Parents/ guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Time to recovery | 3 to 28 days
  Recovery is defined as symptom resolution, exercise tolerance, and normal clinical examination.

SECONDARY OUTCOMES:
Persistence of post-concussive symptoms | 29 to 112 days

CONTACTS AND LOCATIONS:
Overall Officials: John Leddy, MD, Principal Investigator — University at Buffalo; Christina Master, MD, Principal Investigator — Children's Hospital of Philadelphia; Rebekah Mannix, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - University at Buffalo, Buffalo, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leddy JJ, Willer B. Use of graded exercise testing in concussion and return-to-activity management. Curr Sports Med Rep. 2013 Nov-Dec;12(6):370-6. doi: 10.1249/JSR.0000000000000008. PMID 24225521
- [Background] Leddy J, Hinds A, Sirica D, Willer B. The Role of Controlled Exercise in Concussion Management. PM R. 2016 Mar;8(3 Suppl):S91-S100. doi: 10.1016/j.pmrj.2015.10.017. PMID 26972272
- [Background] Leddy JJ, Kozlowski K, Donnelly JP, Pendergast DR, Epstein LH, Willer B. A preliminary study of subsymptom threshold exercise training for refractory post-concussion syndrome. Clin J Sport Med. 2010 Jan;20(1):21-7. doi: 10.1097/JSM.0b013e3181c6c22c. PMID 20051730
- [Background] Leddy JJ, Hinds AL, Miecznikowski J, Darling S, Matuszak J, Baker JG, Picano J, Willer B. Safety and Prognostic Utility of Provocative Exercise Testing in Acutely Concussed Adolescents: A Randomized Trial. Clin J Sport Med. 2018 Jan;28(1):13-20. doi: 10.1097/JSM.0000000000000431. PMID 29257777
- [Derived] Stavisky CJ, Miecznikowski JC, Haider MN, Chizuk HM, Nazir MSZ, Grady MF, McPherson JI, Nowak AS, Willer BS, Master CL, Leddy JJ. Association of Cognitive Symptoms and Abnormal Oculomotor Signs With Recovery in Adolescents After Sport-Related Concussion. Clin J Sport Med. 2025 Mar 1;35(2):138-144. doi: 10.1097/JSM.0000000000001322. Epub 2024 Dec 17. PMID 39692552
- [Derived] Vernau BT, Haider MN, Fleming A, Leddy JJ, Willer BS, Storey EP, Grady MF, Mannix R, Meehan W, Master CL. Exercise-Induced Vision Dysfunction Early After Sport-Related Concussion Is Associated With Persistent Postconcussive Symptoms. Clin J Sport Med. 2023 Jul 1;33(4):388-394. doi: 10.1097/JSM.0000000000001145. Epub 2023 Mar 30. PMID 37015066
- [Derived] Chizuk HM, Willer BS, Cunningham A, Bezherano I, Storey E, Master C, Mannix R, Wiebe DJ, Grady MF, Meehan WP, Leddy JJ, Haider MN. Adolescents with Sport-Related Concussion Who Adhere to Aerobic Exercise Prescriptions Recover Faster. Med Sci Sports Exerc. 2022 Sep 1;54(9):1410-1416. doi: 10.1249/MSS.0000000000002952. Epub 2022 Apr 28. PMID 35482774
- [Derived] Leddy JJ, Master CL, Mannix R, Wiebe DJ, Grady MF, Meehan WP, Storey EP, Vernau BT, Brown NJ, Hunt D, Mohammed F, Mallon A, Rownd K, Arbogast KB, Cunningham A, Haider MN, Mayer AR, Willer BS. Early targeted heart rate aerobic exercise versus placebo stretching for sport-related concussion in adolescents: a randomised controlled trial. Lancet Child Adolesc Health. 2021 Nov;5(11):792-799. doi: 10.1016/S2352-4642(21)00267-4. Epub 2021 Oct 1. PMID 34600629